CLINICAL TRIAL: NCT02935946
Title: Cold Liquids Fed to Preterm Infants: Efficacy and Safety After 10 Minutes of Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Adelphi University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-00901
Record Dates: First submitted 2016-10-13; First posted 2016-10-18 (Estimated); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Deglutition Disorders; Respiratory Aspiration
Keywords: pharyngeal swallow, NICU, intervention, thickening
MeSH Terms: conditions — Deglutition Disorders; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Room Temperature Swallows (No Intervention): Once consented, each participant underwent a video fluoroscopic swallow study (VFSS). Each participant was fed room temperature thin liquid barium (Varibar® Thin Liquid Barium Sulfate for Suspension) from a standard bottle (60ml Similac® Volu-Feeder®) with an attached Similac® Infant Nipple and Ring. The swallows were assessed in real time for any swallowing dysfunction and saved electronically. These swallows were labeled "RTS" for "room temperature swallows. If no swallow dysfunction was observed, the participant became ineligible and the study ended. If swallow dysfunction was observed, the participant became eligible to complete the other arms of the study.
- Cold Liquid Swallows- 5 (Experimental): Immediately following the RTS condition, a total of 5 swallows of Cold Liquid Barium was observed under fluoroscopy from an identical bottle and nipple. Images were saved electronically and labeled "CS5" for "cold swallows-5."
  Interventions: Other: Cold Liquid Barium
- Cold Liquid Swallows- 10 (Experimental): After 10 minutes of feeding a cold liquid, a total of 10 swallows of Cold Liquid Barium was observed under fluoroscopy from an identical bottle and nipple. Images were saved electronically and labeled "CS10" for "cold swallows-10."
  Interventions: Other: Cold Liquid Barium

INTERVENTIONS:
Other: Cold Liquid Barium — Cold Liquid is defined as being between 4-9 °C. One liter bottles of Poland Spring Natural Spring Water will be kept in the radiology suite to remain at room temperature. As described by Fink and colleagues,(42) the bottled water will be used to mix the barium powder to create a thin liquid consistency, with 50% dilution, which is found to be most similar to human milk and infant formula. After the barium is prepared, 2oz will be poured into a bottle and placed in a refrigerator set to 36°F; this will allow the barium to cool to approximately 4-9°C. Before oral administration, the barium mixture will be measured with a thermometer (TP3001 Digital Thermometer from Red Lantern®) to document the exact temperature.
  Arms: Cold Liquid Swallows- 10; Cold Liquid Swallows- 5

SUMMARY:
A previous study revealed that dysphagia preterm infants show statistically significant improvements in their swallowing mechanism when fed cold liquid barium when compared to room temperature liquid barium. The previous study was the first to identify these positive effects, although, only assessed 5 cold liquid swallows, immediately after the room temperature condition. This limited data set restricts the efficacy and safety of using cold liquids in clinical practice, emphasizing the need for further information. The present study aims to objectively assess the influence of cold liquid on the pharyngeal swallow mechanism in preterm infants with dysphagia after 10 minutes of a cold liquid feeding. The investigators will utilize videofluoroscopic swallow studies (VFSS) to analyze the frequency and severity of pharyngeal swallowing deficits during room temperature swallows and compare it to cold liquid swallows at various time points within a 10 minute feeding. Safety measures will also be obtained, such as participant axillary body temperature and gastric content temperature, to identify indicators for the development of cold stress.

DETAILED DESCRIPTION:
Swallowing dysfunction, medically defined as dysphagia, commonly occurs in infants born prematurely due to inadequate timing and coordination of the sensorimotor sequences required for safe swallowing. Approximately 70% of prematurely born infants will be diagnosed with oral, pharyngeal and/or esophageal phase dysphagia with an inverse relationship between severity and gestational age at birth.(1)

Swallowing is extremely important for the infant and child to meet the nutritional requirements for growth and development. When swallowing is dysfunctional, the consequences can be devastating for the infant, possibly resulting morbidity, with complications including pneumonia, respiratory disease, growth compromise or failure to thrive.(1-6) The implications of swallowing difficulty are, therefore, of considerable medical importance to the medical team working with these infants.

A videofluoroscopic swallow study (VFSS) is a widely used assessment for the diagnosis of neonatal dysphagia. VFSS is a definitive investigation to objectively assess the adequacy of airway protection during swallowing and allows simultaneous viewing of the bolus as it passes through the oral, pharyngeal and esophageal stages of swallowing.(7) For infants feeding from a bottle, the clinician relies on the VFSS to both identify and correct the swallowing dysfunction. Several therapeutic techniques or modifications are used during a VFSS to improve swallowing safety in infants, such as various nipple flow rates,(8,9) feeding positions,(10) or pacing the infant's sucking bursts.(11) The most frequently used modification is to thicken the infant's formula or breastmilk to a thicker consistency,(12-14) however, thickening causes some difficulty making it an undesirable option for young infants treated in the neonatal intensive care unit (NICU).(15) These difficulties have resulted in clinicians using alternate therapeutic techniques to treat dysphagia neonates. One alternate technique is to feed the infant cold liquids to stimulate a safer swallow.(16-20)

Original findings obtained by these investigators was the first to indicate that cold liquid swallows reduce airway compromise in dysphagic preterm infants when compared to room temperature liquid. Specifically, the occurrence of deep penetration (p=0.029), aspiration (0.017), mild penetration (p=0.044) and nasopharyngeal reflux (p=0.006) decreased significantly in the cold swallow (CS) condition when compared to the room temperature swallow (RTS) condition during VFSS. Similar findings are documented in adults with dysphagia.(21-35) These positive effects are theorized to occur due to the cold liquid providing the sensory receptors within the pharynx increased sensory information which triggers more efficient swallowing movements.(12,13,21-23)

The original study assessed 5 cold liquid swallows, which provided important information regarding the immediate effects of cold liquids on the pharyngeal swallowing mechanism in preterm infants with dysphagia. Further information regarding the duration of these positive effects is necessary to prove its reliability as a modification to be used at bedside. This study is designed to assess the swallowing mechanism of dysphagic preterm infants after feeding cold liquids for 10 minutes to objectively identify any changes over time.

In addition to the paucity of evidence regarding improved swallowing function over time, the safety of feeding cold liquids remains questionable in the preterm infant population. The greatest concern for these infants is the development of cold stress or altered digestive functioning due to the cold temperature of the liquid. The effects of cold stress in infants are observed in all body systems, including cool skin, tachypnea, respiratory distress, desaturation, increasing episodes of apnea and bradycardia, increased gastric residuals, and emesis.(36) Several older studies have assessed the effects of cold feeds in healthy term and healthy pre term infants, however, study populations may not be representative of todays preterm infant population due to significant medical advances and increased survival rates of extremely preterm infants.

Holt and colleagues(37) found no difference in sleep pattern, vocalizations, motility, intake, feeding behavior, weight gain, temperature or regurgitation in preterm infants with a weight of >1,500gm, when fed cold formula. Gonzalez and colleagues(38) found no significant differences in axillary temperature or gastric residuals in preterm infants fed cold (0-4°C) verses room temperature (25°C) milk. Participants included 14 preterm infants with a gestational age at birth (GAB) of 28-30w, and a mean corrected gestational age of 32 weeks. Anderson and Berseth(39) found no differences in infants' antral or duodenal motor activity as assessed via manometry, as well as gastric emptying among cold (6°C), room temperature (24°C), or body temperature (37°C) feeding groups. This study included preterm infants with GAB 25-36weeks, mean birth weights 915-2,455g. Corrected gestational age of 32-36 weeks at the time of the study. Feedings were given in random order for 3 liquid temperatures. Across all temperatures they found that all infants emptied approximately one third of the bolus feeding by 20 minutes. And across all temperatures approximately 10-20% of the bolus feeding remained in their stomach 2 hours post-prandially. The authors propose that thermo-receptors within the gastrointestinal tract do not appear to be functional in this age group.

Blumenthal and colleagues(40) found no statistical differences between stomach emptying rate in cold (0-4°C), room temperature (25°C) or body temperature (37°C) formula in 20 healthy preterm infants with a mean birth weight of 2.75 ± 0-18 (range 1.49-3.38) kg, and gestation 37-7 ± 0.6 (range 34-41) weeks. They also reported that in all infants the cold feeds were well tolerated and produced no obvious clinical effects.

To assess the potential risks of cold stress, each participant's body temperature will be obtained pre and post cold liquid exposure. To assess digestive functioning, the temperature of each participant's gastric contents will be obtained pre and post cold liquid exposure by extraction of the gastric content via a naso-gastric tube (NGT). If the child does not have a naso-gastric tube in place at the time of the study, the subjects will be enrolled but no documentation of the stomach content temperature will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Infants born prematurely, as defined by birth at less than 37 weeks gestational age, referred for a videofluoroscopic swallow study (VFSS) due to suspected pharyngeal phase dysphagia.

Exclusion Criteria:

* Infants born prematurely with a corrected gestational age of 43 weeks or greater.

Ages: 36 Weeks to 43 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4043 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2024-03-17 (Actual); Study Completion 2024-03-17 (Actual)

PRIMARY OUTCOMES:
Pharyngeal Phase Dysphagia | <5 seconds post swallow trigger
  presence of atypical or disordered movements during the pharyngeal phase of swallowing

SECONDARY OUTCOMES:
Tracheal Aspiration | <5 seconds post swallow trigger
  the occurrence of barium below the level of the true vocal cords
Laryngeal Penetration | <2 seconds post swallow trigger
  the occurrence of barium underneath the epiglottis, in the laryngeal vestibule to the level of the vocal folds
Nasopharyngeal Reflux | <2 seconds post swallow trigger
  the occurrence of barium detected in the nasopharynx, posterior or superior to the velum
Pharyngeal residue | <5 seconds post swallow trigger
  the presence of residual barium coating the pharyngeal walls, pooling in the vallecula or pyriform sinuses post swallow (absent/mild/severe).

CONTACTS AND LOCATIONS:
Overall Officials: Nazeeh Hanna, MD, Principal Investigator — NYU Winthrop Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
in publication

REFERENCES:
- [Background] Newman LA, Keckley C, Petersen MC, Hamner A. Swallowing function and medical diagnoses in infants suspected of Dysphagia. Pediatrics. 2001 Dec;108(6):E106. doi: 10.1542/peds.108.6.e106. PMID 11731633
- [Background] Boesch RP, Wood, RE. (2012). Aspiration. In: Kendig and Chernick's Disorders of the Respiratory Track in Children 8th Edition. Elsevier: Philladelphi: PA, 2012, pp 947-948.
- [Background] Taniguchi MH, Moyer RS. Assessment of risk factors for pneumonia in dysphagic children: significance of videofluoroscopic swallowing evaluation. Dev Med Child Neurol. 1994 Jun;36(6):495-502. doi: 10.1111/j.1469-8749.1994.tb11879.x. PMID 8005360
- [Background] Orenstein SR. Oral, pharyngeal, and esophageal motor disorders in infants and children. GI Motility Online 2006. doi:10.1038/gimo38. Available at: http://www.nature.com/gimo/contents/pt1/full/gimo38.html
- [Background] Smith CH, Logemann JA, Colangelo LA, Rademaker AW, Pauloski BR. Incidence and patient characteristics associated with silent aspiration in the acute care setting. Dysphagia. 1999 Winter;14(1):1-7. doi: 10.1007/PL00009579. PMID 9828268
- [Background] Tutor JD, Gosa MM. Dysphagia and aspiration in children. Pediatr Pulmonol. 2012 Apr;47(4):321-37. doi: 10.1002/ppul.21576. Epub 2011 Oct 18. PMID 22009835
- [Background] Hiorns MP, Ryan MM. Current practice in paediatric videofluoroscopy. Pediatr Radiol. 2006 Sep;36(9):911-9. doi: 10.1007/s00247-006-0124-3. Epub 2006 Mar 22. PMID 16552584
- [Background] Mathew OP. Breathing patterns of preterm infants during bottle feeding: role of milk flow. J Pediatr. 1991 Dec;119(6):960-5. doi: 10.1016/s0022-3476(05)83056-2. PMID 1960618
- [Background] Chang YJ, Lin CP, Lin YJ, Lin CH. Effects of single-hole and cross-cut nipple units on feeding efficiency and physiological parameters in premature infants. J Nurs Res. 2007 Sep;15(3):215-23. doi: 10.1097/01.jnr.0000387617.72435.c6. PMID 17806038
- [Background] Clark L, Kennedy G, Pring T, Hird M. Improving bottle feeding in preterm infants: Investigating the elevated side-lying position. Infant 2007; 3:154-158.
- [Background] Law-Morstatt L, Judd DM, Snyder P, Baier RJ, Dhanireddy R. Pacing as a treatment technique for transitional sucking patterns. J Perinatol. 2003 Sep;23(6):483-8. doi: 10.1038/sj.jp.7210976. PMID 13679936
- [Background] Logemann JA. The dysphagia diagnostic procedure as a treatment efficacy trial. Clin Commun Disord. 1993 Fall;3(4):1-10. PMID 8111359
- [Background] Ruark JL, McCullough GH, Peters RL, Moore CA. Bolus consistency and swallowing in children and adults. Dysphagia. 2002 Winter;17(1):24-33. doi: 10.1007/s00455-001-0098-0. PMID 11820384
- [Background] Khoshoo V, Ross G, Kelly B, Edell D, Brown S. Benefits of thickened feeds in previously healthy infants with respiratory syncytial viral bronchiolitis. Pediatr Pulmonol. 2001 Apr;31(4):301-2. doi: 10.1002/ppul.1043. PMID 11288213
- [Background] Cichero JA, Nicholson TM, September C. Thickened milk for the management of feeding and swallowing issues in infants: a call for interdisciplinary professional guidelines. J Hum Lact. 2013 May;29(2):132-5. doi: 10.1177/0890334413480561. Epub 2013 Mar 18. No abstract available. PMID 23507962
- [Background] Arvedson JC & Lefton-Greif MA. 1998. Pediatric Videofluoroscopic Swallow Studies: A Professional Manual with Caregiver Guidelines. San Antonio, TX: Communication Skill Builders, Division of Psychologic Corp, Harcourt Assessment, Inc. Available at www.PsychCorp.com.
- [Background] Fraker C & Walbert L. Evaluation and Treatment of Pediatric Feeding Disorders: From NICU to Childhood. Pro-Ed: Austin TX, 2003.
- [Background] Swigert N. Source for pediatric dysphagia. Singular: San Diego, CA, 1998.
- [Background] Wolf LS & Glass RP. Feeding and Swallowing Disorders in Infancy: Assessment and Management. Therapy Skill Builders: Tucson, AZ, 1992.
- [Background] Arvedson JC & Brodsky L. Pediatric Swallowing and Feeding: Assessment and Management. Singular Publishing Group: Albany, NY, 2002.
- [Background] Dantas RO, Kern MK, Massey BT, Dodds WJ, Kahrilas PJ, Brasseur JG, Cook IJ, Lang IM. Effect of swallowed bolus variables on oral and pharyngeal phases of swallowing. Am J Physiol. 1990 May;258(5 Pt 1):G675-81. doi: 10.1152/ajpgi.1990.258.5.G675. PMID 2333995
- [Background] Bisch EM, Logemann JA, Rademaker AW, Kahrilas PJ, Lazarus CL. Pharyngeal effects of bolus volume, viscosity, and temperature in patients with dysphagia resulting from neurologic impairment and in normal subjects. J Speech Hear Res. 1994 Oct;37(5):1041-59. doi: 10.1044/jshr.3705.1041. PMID 7823550
- [Background] Ebihara S, Kohzuki M, Sumi Y, Ebihara T. Sensory stimulation to improve swallowing reflex and prevent aspiration pneumonia in elderly dysphagic people. J Pharmacol Sci. 2011;115(2):99-104. doi: 10.1254/jphs.10r05cp. Epub 2011 Jan 18. PMID 21258172
- [Background] Teismann IK, Steinstrater O, Warnecke T, Suntrup S, Ringelstein EB, Pantev C, Dziewas R. Tactile thermal oral stimulation increases the cortical representation of swallowing. BMC Neurosci. 2009 Jun 30;10:71. doi: 10.1186/1471-2202-10-71. PMID 19566955
- [Background] Miura Y, Morita Y, Koizumi H, Shingai T. Effects of taste solutions, carbonation, and cold stimulus on the power frequency content of swallowing submental surface electromyography. Chem Senses. 2009 May;34(4):325-31. doi: 10.1093/chemse/bjp005. Epub 2009 Feb 16. PMID 19221127
- [Background] Miyaoka Y, Haishima K, Takagi M, Haishima H, Asari J, Yamada Y. Influences of thermal and gustatory characteristics on sensory and motor aspects of swallowing. Dysphagia. 2006 Jan;21(1):38-48. doi: 10.1007/s00455-005-9003-6. PMID 16544093
- [Background] Regan J, Walshe M, Tobin WO. Immediate effects of thermal-tactile stimulation on timing of swallow in idiopathic Parkinson's disease. Dysphagia. 2010 Sep;25(3):207-15. doi: 10.1007/s00455-009-9244-x. Epub 2009 Aug 26. PMID 19707818
- [Background] Lazzara G, Lazarus C, Logemann JA. Impact of thermal stimulation on the triggering of the swallowing reflex. Dysphagia 1986; 1(2): 73-77.
- [Background] Cola PC, Gatto AR, Silva RG, Spadotto AA, Schelp AO, Henry MA. The influence of sour taste and cold temperature in pharyngeal transit duration in patients with stroke. Arq Gastroenterol. 2010 Jan-Mar;47(1):18-21. doi: 10.1590/s0004-28032010000100004. PMID 20520970
- [Background] Hamdy S, Jilani S, Price V, Parker C, Hall N, Power M. Modulation of human swallowing behaviour by thermal and chemical stimulation in health and after brain injury. Neurogastroenterol Motil. 2003 Feb;15(1):69-77. doi: 10.1046/j.1365-2982.2003.00390.x. PMID 12588471
- [Background] Selcuk B, Uysal H, Aydogdu I, Akyuz M, Ertekin C. Effect of temperature on electrophysiological parameters of swallowing. J Rehabil Res Dev. 2007;44(3):373-80. doi: 10.1682/jrrd.2006.08.0089. PMID 18247234
- [Background] Rosenbek JC, Robbins J, Fishback B, Levine RL. Effects of thermal application on dysphagia after stroke. J Speech Hear Res. 1991 Dec;34(6):1257-68. doi: 10.1044/jshr.3406.1257. PMID 1787707
- [Background] Selinger M, Prescott TE, McKinley R. The efficacy of thermal stimulation: A case study. Rocky Mountain J Commun Disord 1990; 6:21-23.
- [Background] Bove M, Mansson I, Eliasson I. Thermal oral-pharyngeal stimulation and elicitation of swallowing. Acta Otolaryngol. 1998 Sep;118(5):728-31. doi: 10.1080/00016489850183269. PMID 9840513
- [Background] Dumm M, Hamms M, Sutton J, Ryan-Wenger N. NICU breast milk warming practices and the physiological effects of breast milk feeding temperatures on preterm infants. Adv Neonatal Care. 2013 Aug;13(4):279-87. doi: 10.1097/ANC.0b013e31829d8c3a. PMID 23912021
- [Background] HOLT LE Jr, DAVIES EA, HASSEL MEYER EG, ADAMS AO. A study of premature infants fed cold formula. J Pediatr. 1962 Oct;61:556-61. doi: 10.1016/s0022-3476(62)80146-2. No abstract available. PMID 13908574
- [Background] Gonzales I, Duryea EJ, Vasquez E, Geraghty N. Effect of enteral feeding temperature on feeding tolerance in preterm infants. Neonatal Netw. 1995 Apr;14(3):39-43. PMID 7603419
- [Background] Anderson CA, Berseth CL. Neither motor responses nor gastric emptying vary in response to formula temperature in preterm infants. Biol Neonate. 1996;70(5):265-70. doi: 10.1159/000244375. PMID 8955912
- [Background] Blumenthal I, Lealman GT, Shoesmith DR. Effect of feed temperature and phototherapy on gastric emptying in the neonate. Arch Dis Child. 1980 Jul;55(7):562-4. doi: 10.1136/adc.55.7.562. PMID 7436507
- [Background] Fink TA, Ross JB. Are we testing a true thin liquid? Dysphagia. 2009 Sep;24(3):285-9. doi: 10.1007/s00455-008-9203-y. Epub 2009 Feb 21. PMID 19234743
- [Background] Lee JH, Chang YS, Yoo HS, Ahn SY, Seo HJ, Choi SH, Jeon GW, Koo SH, Hwang JH, Park WS. Swallowing dysfunction in very low birth weight infants with oral feeding desaturation. World J Pediatr. 2011 Nov;7(4):337-43. doi: 10.1007/s12519-011-0281-9. Epub 2011 Oct 20. PMID 22015726
- [Background] Mercado-Deane MG, Burton EM, Harlow SA, Glover AS, Deane DA, Guill MF, Hudson V. Swallowing dysfunction in infants less than 1 year of age. Pediatr Radiol. 2001 Jun;31(6):423-8. doi: 10.1007/s002470100456. PMID 11436889
- [Background] Weir KA, McMahon SM, Long G, Bunch JA, Pandeya N, Coakley KS, Chang AB. Radiation doses to children during modified barium swallow studies. Pediatr Radiol. 2007 Mar;37(3):283-90. doi: 10.1007/s00247-006-0397-6. Epub 2007 Jan 10. PMID 17216172
- [Background] The Alliance for Radiation Safety in Pediatric Imaging. FAQ. http://www.pedrad.org/associations/5364/ig/ index.cfm?page=669. Accessed on February 20, 2013.